CLINICAL TRIAL: NCT01748838
Title: A Phase I Randomised, Double-Blind, Placebo-Controlled, Ascending Single & Repeat-Dose Study of Safety, Tolerability & Pharmacokinetics of CTX-4430 When Administered Orally to Healthy Adult Subjects
Brief Title: Phase 1 Study Assessing the Safety and Tolerability of CTX-4430
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celtaxsys, Inc. (Other)
Collaborators: Clinical Network Services (Unknown); Linear Clinical Research (Industry); CPR Pharma Services Pty Ltd, Australia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTX-4430-HV-001
Record Dates: First submitted 2012-12-08; First posted 2012-12-13 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Pulmonary Inflammation
MeSH Terms: conditions — Pneumonia | interventions — acebilustat; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part 1: CTX-4430 (Experimental)
  Interventions: Drug: CTX-4430; Other: Mannitol
- Part 1: Placebo + Mannitol (Placebo Comparator)
  Interventions: Other: Mannitol; Drug: Placebo
- Part 2: CTX-4430 (Experimental)
  Interventions: Drug: CTX-4430; Other: Mannitol
- Part 2: Placebo + Mannitol (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Mannitol

INTERVENTIONS:
Drug: CTX-4430 — Ascending single oral doses of CTX-4430 will be administered to subjects in 6 cohorts on day 1. Following a 14-day washout, subjects in two of the six cohorts will cross-over, fed a high fat diet and administered different single oral doses of CTX-4430
  Arms: Part 1: CTX-4430
Other: Mannitol — excipient blended with CTX-4430 in capsules
  Other Names: osmitrol
  Arms: Part 1: CTX-4430; Part 1: Placebo + Mannitol
Drug: Placebo — Single oral doses of placebo will be administered to subjects in 6 cohorts on day 1. Following a 14-day washout, subjects in two of the six cohorts will cross over, fed a high fat diet and administered single oral doses of placebo
  Arms: Part 1: Placebo + Mannitol
Drug: CTX-4430 — Ascending repeat doses of CTX-4430 will be administered orally, once-daily, to subjects in 4 cohorts on days 1-14.
  Arms: Part 2: CTX-4430
Drug: Placebo — Repeat doses of placebo will be administered orally, once-daily, to subjects in 4 cohorts on days 1-14.
  Arms: Part 2: Placebo + Mannitol
Other: Mannitol — excipient blended with CTX-4430
  Other Names: osmitrol
  Arms: Part 2: CTX-4430; Part 2: Placebo + Mannitol

SUMMARY:
The purpose of this study is to assess the safety and tolerability of CTX-4430 capsules taken orally once daily in normal healthy volunteers. CTX-4430 is being developed to treat lung inflammation that occurs in cystic fibrosis (CF). This study includes two-parts: Part 1 assesses single dosing; and Part 2 assesses repeat dosing for 14 days. Each part will include several dosages. During the single-dose part of the study, following a 14-day washout period, two cohorts will be assessed for potential effects on tolerability when fed at the time of dosing. For both parts of the study, blood samples will be collected for PK assay validation.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, 18 to 55 years of age
* Medically healthy
* Body mass index ≥ 18.0 and ≤ 29.9
* Non-tobacco/nicotine-containing product users 6 months prior to the first study drug administration
* Negative urine drug/alcohol screen prior to Day -1
* Voluntary consent
* Male agrees to be sexually abstinent or to use a condom when engaging in sexual activity through completion
* Females of childbearing potential must either be sexually inactive for 14 days prior to the first study drug administration and remain so through 30 days following the final dosing of the study drug, or have been using one of the following methods of birth control for the times specified:
* Intra-uterine device in place for at least 3 months prior
* Double barrier method for at least 14 days prior
* Male partner who is surgical sterile at least 6 months prior to first study drug administration and is sole sexual partner for that female
* Adequate hormonal contraception.Female subjects who become sexually active during the course of the study must use a double barrier method from the start of sexual activity through 30 days following the final dosing
* Females of non-childbearing potential have undergone one of the following sterilization procedures at least 6 months prior to first study drug administration:
* Essure® sterilization and be using a barrier method throughout the study
* bilateral tubal ligation with a barrier method throughout the study
* hysterectomy
* bilateral oophorectomy or be postmenopausal with amenorrhea for at least 1 year prior to the first study drug administration and follicle stimulating hormone serum levels ≥40 mIU/mL
* Subject has a Forced Expiratory Volume of ≥80% of predicted at screening
* Subject has a resting oxygen saturation >92% on room air

Exclusion Criteria:

* Positive testing for human immunodeficiency virus,hepatitis B surface antigen, or hepatitis C antibodies
* Subject is febrile at any stage from screening until pre-dose
* History or presence of alcoholism or drug abuse within 2 years prior to the first study drug administration
* Hypersensitivity or idiosyncratic reaction to compounds related to CTX-4430.
* Use of any over-the-counter medication,(including herbal products and vitamin supplements),within the 7 days prior to the Day 1. Use of any nonsteroidal anti-inflammatory drugs,aspirin,antirheumatic drugs, leukotriene receptor antagonists, leukotriene enzyme inhibitors within the 14 days prior to the first study drug administration or 5 half-lives,whichever is longer. Administration or use of oral,inhaled, intranasal, parenteral, or >1% topical glucocorticoids within the 6 months prior to Day 1
* Use of any significant inhibitors or substrates of OAT3, OCT2 and/or OATP P1/B1 within 30 days prior to the first study drug administration
* Blood donation or significant blood loss within 60 days prior to the first study drug administration
* Plasma donation within 7 days prior to the first study drug administration.
* Participation in another clinical trial within 30 days prior to the first study drug administration
* Females who are pregnant or lactating
* Clinically relevant surgery within the past three months prior to first drug administration
* Personal or family history of prolonged QT syndrome; or a QTc interval >430 msec (males) or >450 msec (females)
* Sitting blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg
* Pulse is higher than 100 b.p.m.
* Regular alcohol consumption in males >21 units per week and females >14 units per week
* Failure to satisfy the PI of fitness to participate for any reason
* Active infection
* History of seizure
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine,immunologic, dermatologic, neurological, or psychiatric disease
* Use of any prescription medication within 14 days prior to Day 1
* Acute illness within 30 days prior to Day 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CTX-4430 in healthy subjects by evaluating changes in physical exams, laboratory tests, vital signs (e.g., blood pressure), pulmonary function tests, ECGs, and the occurrence and severity of adverse events. | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Janakan Krishnarajah, MB, BS FRACP, Principal Investigator — Linear Clinical Research
Locations (1):
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia